CLINICAL TRIAL: NCT01730885
Title: A Trial Investigating the Accuracy and Precision of the BGStar® and iBGStar® Blood Glucose Meter in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: BGStar
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BGStar (Other): Comparision
  Interventions: Other: Comparison of different Blood Glucose Meters

INTERVENTIONS:
Other: Comparison of different Blood Glucose Meters

SUMMARY:
Due to continuing technological progress and better understanding of the needs for glucose monitoring, the performance requirements of blood glucose meters, primarily regarding their accuracy, are constantly debated and keep evolving as a consequence. Recently a discussion was initiated by the Food and Drug Administration (FDA) to improve the accuracy of BG meters in the point-of-care testing setting by asking for fulfilment of higher requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
2. Male or female subjects aged 18-74 years (both inclusive).
3. Type 1 diabetes mellitus (as diagnosed clinically) ≥ 12 months.
4. Body mass index 18.0-28.0 kg/m2 (both inclusive).
5. HbA1c ≤ 9.0 % by local laboratory analysis.

Exclusion Criteria:

1. Known or suspected hypersensitivity to lancet fingerpricks / needle injections.
2. Previous participation in this trial. Participation is defined as having performed at least one BG meter measurement as part of the study.
3. Receipt of any investigational medicinal product within 30 days before randomisation in this trial.
4. Formation of callus on the fingertips or any other skin condition that may hamper fingerprick blood sampling and/or insufficient capillary blood volume sampling (< 50 μL) during test fingerprick(s).
5. Haemoglobin < 8.0 mmol/L (male) or < 6.4 mmol/L (female), total leukocyte count < 3.0 x 109/L, thrombocytes <100 x 109/L, serum creatinine levels ≥ 126 μmol/L (male) or ≥ 111 μmol/L (female), bilirubin > 3x the upper limit of normal (ULN), and alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and gamma-glutamyl transferase (γ-GT) > 2 x ULN.
6. Suffer from or history of a life threatening disease (i.e. cancer except basal cell skin cancer or squamous cell skin cancer), or any clinically significant respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (with the exception of diabetes mellitus and euthyroid struma), haematological, dermatological, venereal, -

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Mean absolute relative deviation (MARD) from paired reference values of BGStar®, iBGStar® and comparator BG meter measurements at stable hypoglycaemic, euglycaemic and hyperglycaemic levels and overal | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany